CLINICAL TRIAL: NCT01893762
Title: Innate Immune Response to Anaerobe and Aerobe Exercise in Rowing Athletes
Brief Title: Innate Immune Response to (An)Aerobic Exercise in Rowing Athletes
Acronym: INCREASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, B. Hilvering, M.D., UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCREASE-2013
Record Dates: First submitted 2013-06-27; First posted 2013-07-09 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Upper Respiratory Tract Infections; URTI
Keywords: neutrophil; exercise; URTI; Innate; Immune
MeSH Terms: conditions — Respiratory Tract Infections; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 16 rowers (Experimental): Adult rowers, aged between 18 and 25, training >6 times a week are subjected to both an aerobic and a an anaerobic exercise challenge. Between the two challenges there must a pause of at least a week.
  Interventions: Biological: Aerobic exercise; Biological: Anaerobic exercise

INTERVENTIONS:
Biological: Aerobic exercise — Aerobic exercise: 2x30 min on an indoor rowing machine at 75% of Maximum heart rate
Biological: Anaerobic exercise — Anaerobic exercise: 3x1000m maximum effort, on an indoor rowing machine

SUMMARY:
Exercise induces innate immune response activation in athletes. The response starts during exercise and lasts for approximately 24 hours. This innate immune response shows similarities to the innate immune activation observed in, for example, bacterial infection and trauma. Immediately after exercise, athletes develop leukocytosis and cytokine production is altered towards an inflammatory pattern. However, to gain insight in immune response, a detailed cell receptor expression is required. To investigate the physiological innate immune response to exercise, we developed a model in rowers.

Aim: To determine the type and degree of cellular inflammatory response in peripheral blood of elite rowing athletes after both anaerobe and aerobe exercise.

Study design:

Investigator driven, monocenter observational pilot study.

Study population: 16 healthy, non-asthmatic, human volunteers, 18-25 year old. All competitive rowing athletes.

DETAILED DESCRIPTION:
Rationale: Exercise induces innate immune response activation in athletes. The response starts during exercise and lasts for approximately 24 hours. This innate immune response shows similarities to the innate immune activation observed in, for example, bacterial infection and trauma. Immediately after exercise, athletes develop leukocytosis and cytokine production is altered towards an inflammatory pattern. However, to gain insight in immune response, a detailed cell receptor expression is required. To investigate the physiological innate immune response to exercise, we developed a model in rowers.

Objective: To determine the type and degree of cellular inflammatory response in peripheral blood of elite rowing athletes after both anaerobe and aerobe exercise.

Study design: Investigator driven, monocenter observational pilot study.

Study population: 16 healthy, non-asthmatic, human volunteers, 18-25 year old. All competitive rowing athletes.

Intervention : All athletes perform two separate tests on a rowing ergometer. One anaerobe (flat out) exercise test (minutes) at day 1 and a aerobe test (1 hour) at day 2. Blood withdrawal of 9mL will be performed at four time points (1 pretest time point and 3 post: at 0h, 2 and 4h).

Main study parameters/endpoints: The main endpoint is a rise in neutrophil cell count and the appearance of different subsets of neutrophils objectified by a change in receptor expression. Not only neutrophils are important in this innate cell response, other leukocytes like lymphocytes, monocytes and hematopoietic progenitor cells also play a role. Therefore the detailed analysis of receptor profiles on these cells will be measured by Flowcytometry.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The anaerobe and aerobe exercise tests do not differ significantly from what the athletes are used to do for training purposes. Athletes who experience any pain or discomfort during exercise will be advised to stop. Blood withdrawal on itself may cause a vasovagal response and especially well trained athletes are susceptible to develop this response. A trained physician is present to take care and look after rowers that suffered from vasovagal collapse. All anaerobe exercise brings along a very small risk of acute cardiovascular complications and although all rowers undergo exercise testing by an exercise physiologist before participating in competition, this risk remains.

The total amount of time of the study is 2 times 5 hours. This time frame consists of the prior blood withdrawal, the testing itself and subsequently the three time points of blood withdrawal. The amount of blood withdrawal per athlete is 4 x 9mL, with a total of 36 mL per volunteer at one day of testing. The total blood withdrawal is therefore 72 mL base on two testing days.

ELIGIBILITY:
Inclusion Criteria:

* Elite rower: rowing for 12 months or longer, >6 times a week.
* Aged 18-25 years
* Pretested(by exercise test*) maximum heart rate
* Visiting Rowing club Triton, Orca or Viking
* Performed a sports medical examination test (required for competing on a national level by the Royal Dutch Rowing Asscociation) *The exercise test is a multi step power test which builds up to maximum effort.

Exclusion Criteria:

* Asthmatic
* Current respiratory infection, sinusitis, otitis or any other sign of acute/ chronic inflammatory disease
* Physically injured

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2013-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in neutrophil surface marker expression profiles over time | pre, 0h, 2h and 4h
  FACS analysis of peripheral blood neutrophils. The changes in surface markers over time will be analysed by principal component analysis.

SECONDARY OUTCOMES:
Functional differences of neutrophil phenotypes before versus neutrophils that appear after exercise | pre and 2h post
  Neutrophils: Oxidative burst, killing capacity of St. Aureus, chemotaxis
Changes in absolute cell count | pre, 0, 2h and 4h
  Measuring the change in absolute cell count (granulocytes, lymphocytes, monocytes) over time. Timepoint 'pre' is considered to be the basal level and 0, 2 and 4h as points of change. Repeated measures ANOVA will be used to detect the change.

OTHER OUTCOMES:
Differences between anaerobic and aerobic exercise in neutrophil surface marker expression, functionality of neutrophils and absolute cell counts (granulocytes, lymphocytes and monocytes) | pre, 0h, 2h, 4h
  Compare the peripheral blood leukocyte characteristics in the context of anaerobic versus aerobic exercise challenge
  * Surface marker expression
  * Functional differences
  * Absolute cell counts

CONTACTS AND LOCATIONS:
Overall Officials: Bart Hilvering, M.D., Study Director — UMC Utrecht, department of Respiratory Medicine; Leo Koenderman, Professor, Principal Investigator — UMC Utrecht, department of Respiratory Medicine; Daan Switters, Study Director — UMC Utrecht
Locations (1):
- Rowing Centre "De Driewerf", Utrecht, Utrecht, Netherlands